CLINICAL TRIAL: NCT04513002
Title: A Phase 2A/2B Placebo-controlled Randomised Clinical Trial to Test the Ability of Triheptanoin to Protect Primary Airway Epithelial Cells Obtained From Participants With Ataxia-telangiectasia Against Death Induced by Glucose Deprivation
Brief Title: Ataxia-telangiectasia: Treating Mitochondrial Dysfunction With a Novel Form of Anaplerosis
Acronym: A-TC7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: A-T2020/01
Record Dates: First submitted 2020-07-26; First posted 2020-08-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2021-11

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia Telangiectasia; Anaplerosis
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — triheptanoin

STUDY DESIGN:
Intervention Model Description: 1. Primary objective A combined phase 2A/B trial will be undertaken to determine optimal dose, demonstrate tolerability, and to examine efficacy and safety of triheptanoin in participants with A-T.
  2. Secondary objectives
     * Determine to what extent the beneficial effects of triheptanoin on epithelial cells in culture translate to clinical efficacy in patients with A-T. Clinical endpoints will include ataxia rating; MRI imaging; lung function; eye movement changes and speech assessment.
     * Provide validation of our primary and secondary endpoints to plan a phase 3 trial and form the basis of future trials.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once all required screening assessments are completed and eligibility is confirmed, participants will be registered with the Sponsor. Upon approval of registration, participants will be assigned a unique participant number that will remain consistent for the duration of the study.
  Participants will be randomised (RandoWeb) into one of the following three groups on a 1:1 ratio:
  1. Group 1: 10%, 20%, 35%, 35%, 35%,35%.
  2. Group 2: placebo, 10%, 20%, 35%, 35%,35%.
  3. Group 3; placebo, placebo, 10%, 20%, 35%,35%.
  Our study pharmacist will ensure the groups are blinded in terms of dose increases, volumes, colour and taste of liquid dispensed in triheptanoin and placebo (medium chain triglyceride oil).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Triheptanoin and no Placebo (Other): Parallel group, placebo-controlled, dose-escalation each 2 months for 12 months. Dose based on percent (%) of calculated caloric intake.
  Thirty participants will be randomised in blocks on a 1:1:1 ratio into one of three groups.
  Group 1: 10%, 20%, 35%, 35%, 35% (no placebo). Group 2: placebo, 10%, 20%, 35%, 35% Group 3: placebo, placebo, 10%, 20%, 35%
  Interventions: Dietary Supplement: Triheptanoin
- Group 2: Placebo and Triheptanoin (Other): Parallel group, placebo-controlled, dose-escalation each 2 months for 12 months. Dose based on percent (%) of calculated caloric intake.
  Thirty participants will be randomised in blocks on a 1:1:1 ratio into one of three groups.
  Group 1: 10%, 20%, 35%, 35%, 35% (no placebo). Group 2: placebo, 10%, 20%, 35%, 35% Group 3: placebo, placebo, 10%, 20%, 35%
  Interventions: Dietary Supplement: Triheptanoin
- Group 3: Placebo, Placebo and Triheptanoin (Other): Parallel group, placebo-controlled, dose-escalation each 2 months for 12 months. Dose based on percent (%) of calculated caloric intake.
  Thirty participants will be randomised in blocks on a 1:1:1 ratio into one of three groups.
  Group 1: 10%, 20%, 35%, 35%, 35% (no placebo). Group 2: placebo, 10%, 20%, 35%, 35% Group 3: placebo, placebo, 10%, 20%, 35%
  Interventions: Dietary Supplement: Triheptanoin

INTERVENTIONS:
Dietary Supplement: Triheptanoin — Triheptanoin is a highly purified, synthetic medium odd-chain triglyceride that is catabolized to heptanoate.

SUMMARY:
Study design: Parallel group, placebo-controlled, dose-escalation each 2 months for 12 months. Dose based on percent (%) of calculated caloric intake. Thirty participants will be randomised in blocks on a 1:1:1 ratio into one of three groups stratified by age (< 5 years, 5-10 years, > 10 years of age). Group 1: 10%, 20%, 35%, 35%, 35% (no placebo). Group 2: placebo, 10%, 20%, 35%, 35% Group 3: placebo, placebo, 10%, 20%, 35%.

Primary endpoint: The percent cell death induced by glucose deprivation in cell culture. Secondary endpoints include: Scales for assessment and rating of ataxia, International Cooperative Ataxia Rating Scale, Ataxia Telangiectasia Neurological Examination Scale Toolkit, speech and language assessment, EyeSeeCam assessment, MRI lung imaging, Lung function, Upper respiratory microbiome, Faecal microbiome, Survival and inflammatory phenotype of airway epithelial cells, macrophages and in serum, Metabolomic biomarker discovery in serum and measurement of neuroflament light chain.

DETAILED DESCRIPTION:
Ataxia Telangiectasia (A-T) is a rare, genetic, progressive, life-limiting, neuro-degenerative condition affecting a variety of body systems resulting in ataxia, immune deficiency, respiratory complications and a predisposition to cancer. Currently there is no cure for A-T. Over the years, a number of small clinical trials using steroids, antioxidants and anti-inflammatory agents have had little success. The disease natural history is relentless leading to early death. A-T generates a significant disease burden for the individuals, their extended families and on health care resources. With palliative care being the only current option for families, a treatment trial for A-T meets an unmet need. The investigators preliminary data provide compelling evidence of reversible mitochondrial dysfunction and preventable cell death in A-T patient cells and the beneficial effects of heptanoate (C7), the primary metabolite of triheptanoin. C7 corrects a defect in endoplasmic reticulum (ER)-mitochondrial signalling in A-T cells and has great potential for application in treating participants. C7 has been utilised with efficacy and safety over the last 15 years for inborn errors of metabolism (IEM) such as long chain fatty acid defects (LC-FAOD).

A-T is due to a genetic defect that results in a defective serine/threonine protein kinase, known as ATM. Normally, ATM, plays a central role in protecting the genome against damage. It is increasingly evident that ATM protects cells against oxidative stress. This protein is also present outside the nucleus, where it is activated by oxidative stress through a separate mechanism from DNA damage, providing an explanation why anti-oxidants have a protective role in A-T cells in culture and in animal models. From these and other studies, it is evident that mitochondrial abnormalities characterise ATM and it has been suggested that A-T should be considered, at least in part, as a mitochondrial disease. The Investigators have added substance to that claim by showing that ATM-deficient (B3) cells are exquisitely sensitive to inhibition of glycolysis by glucose deprivation, compared to controls (HBEC). The investigators have also shown this increased sensitivity to nutrient deprivation for primary epithelial cells from patients and in immortalised patient cells. Together these data point to a reduced capacity of A-T mitochondria to support energy metabolism and provide additional evidence for a mitochondrial defect in A-T cells. The investigators have recently demonstrated that this hypersensitivity to glucose deprivation can be explained by a novel mechanism involving defective signalling between the ER and the mitochondrion. The investigators demonstrated that this was caused by defective assembly of the VDAC1-GRP75-IP3R1 calcium channel and less ER-mitochondria contact points as determined by transmission electron microscopy. This in turn resulted in reduced calcium release from the ER and less transfer to mitochondria providing further evidence for mitochondrial dysfunction in A-T cells.

The investigators selected triheptanoin, a highly purified, synthetic medium odd-chain triglyceride that is catabolized to heptanoate and can traverse the mitochondrial membrane without the carnitine carrier. Free heptanoate is then metabolized by the medium chain fatty acid oxidation enzymes to yield both acetyl CoA and propionyl CoA that act as anaplerotics to replenish the TCA cycle and enhance energy metabolism by providing NADPH and generating ATP. The investigators demonstrated that heptanoate partially corrects the extreme sensitivity to glycolysis inhibition in both the ATM-deficient cell line as well as in primary epithelial cells from a patient with A-T. Excitingly, heptanoate also corrected all of the defects in ER-mitochondrial signalling including calcium uptake into mitochondria. Based on the importance of mitochondrial dysfunction in the A-T phenotype and our results revealing correction of mitochondrial function by heptanoate, the investigators consider that triheptanoin has excellent potential in correcting many aspects of the A-T phenotype including the progressive neurodegenerative phenotype.

Triheptanoin has been used for over 15 years to treat LC-FAOD, with demonstrated improvements in cardiac function and reductions in rhabdomyolysis episodes. Triheptanoin and heptanoate are known to protect against cell death in experimental conditions largely characterised by oxidative stress, such as stroke and motor neurone disease, adult polyglucosan body disease, alternating hemiplegia of childhood, Glucose-1 transporter deficiency, and mouse models and humans with epilepsy. Heptanoate protects cultured neurons against H2O2-induced cell death. Collectively these studies demonstrate that triheptanoin is well tolerated and is effective in treating a range of neurological conditions associated with neuronal energy deficiency.

Seamless Phase II to Phase III go/no-go criteria Interim monitoring for the intervention program in the A-T2020/01 trial will occur at the times of the two interim analyses (first, when the study cohort has completed the initial 2 months treatment, and second, after 6 months treatment when Group One has completed 2 months of the 35% dose). A blinded report will be presented to the iDSMB containing pertinent descriptive statistics of the groups, a standard between-group comparison for the primary and secondary outcomes, and a Bayesian estimation of the (posterior) probability that each of the three intervention groups is superior for the primary outcomes. The information to be presented to the iDSMB will be agreed with the iDSMB prior to the first iDSMB meeting, and will be updated at the time of the iDSMB meetings. Data will be presented to the iDSMB in a blind fashion, but the iDSMB can request unblinded data to confirm or ratify any reported interim results. The iDSMB may however make a recommendation about stopping current interventions if they show poor promise or futility.

The primary endpoints for interim iDSMB reports are the percent cell death induced by glucose deprivation in cell culture, and reversal/correction of their abnormal mitochondrial profile in primary epithelial cells resulting in cell death over the treatment period.

Secondary scales clinical neurological assessments assist formulating the go/no-go criteria and will include: SARA and ICARS. SARA is a validated cerebellar ataxia tool, measuring gait, stance, sitting, speech, finger-chase test, finger nose-test, fast alternating movements and heel-shin test. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia); Gait (0-8 points), Stance (0-6 points), Sitting (0-4 points), Speech disturbance (0-6 points), Finger chase (0-4 points), Nose-finger test (0-4 points), Fast alternating hand movement (0-4 points), Heel-shin slide (0-4 points). ICARS is a scale recorded out of 100 with 19 items and 4 subscales and has been used in A-T. Disorders rated as subscales within the ICARS are: Postural and gait disturbances, (7 items, 0-34 points) Limb Ataxia (7 items, 0-52 points), Dysarthria (2 items, 0-8 points), and Oculomotor disorders (3 items, 0-6 points). Minimum Score: 0 Maximum score: 100.

go/no-go triggers

go triggers Seamless progress from Phase II to Phase III will be triggered under the following pre-set parameters;

* If clinically or statistically significant improvement in the primary study outcome is observed in combination with a measured improvement of at least ½ standard deviation in key clinical scales which includes either;
* significant improvement in total combined scores from the SARA and ICARS scales.
* And/or significant improvements any aspects of the SARA and ICARS scales individually, especially pertaining to; Postural and gait improvements, Speech disturbance, Improved fine motor skills, Fine motor disturbance, Kinetic functions

No-go triggers Seamless progress from Phase II to Phase III will not occur under the following pre-set parameters;

* Adverse events
* If no clinically significant improvement in the primary study outcome is observed
* If a clinically significant improvement in the primary study outcome occurs without any improvements in key secondary scales specifically the SARA and ICARS.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, of any age, with a confirmed diagnosis of A-T,
* Patients who are able to undertake the study procedures,
* Families who are able to comply with the protocol for its duration and who provide informed patient assent and consent signed and dated by parent/legal guardian or adult participant according to local regulations.

Exclusion Criteria:

* Patients whose parents/legal guardians are not able to provide consent
* Patients who have been in another randomised clinical intervention trial where the use of investigational medicinal product within 3 months or 5 half-lives, whichever is longer, before study enrolment
* Taking off label mediations or nutritional supplements that the PI consider would impact participant's safe participation.
* Patients who are pregnant and/or lactating, planning a pregnancy during the study. Contraception must be used for sexually active male and female participants
* Intestinal Malabsorption secondary to Pancreatic Insufficiency
* Liver enzymes (alanine aminotransferase [ALT]/aspartate aminotransferase [AST]) or total bilirubin > 2 x the upper limit of normal at the time of screening.
* Renal insufficiency as defined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 at the screening visit.
* Any comorbid medical condition that in the assessment of the PI that would impact participant's safe participation (e.g. active cancer requiring treatment)
* Evidence of dysphagia that places subject at risk of aspiration if orally fed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 1, baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 60, assessment of effects/changes from Day 1 baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 120, assessment of effects/changes from Day 60 baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 180, assessment of effects/changes from Day 120 baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 240, assessment of effects/changes from Day 180 baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 300, assessment of effects/changes from Day 240 baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.
Nasal epithelial cell survival under conditions of glucose deprivation. | Day 360, assessment of effects/changes from Day 300 baseline measurement
  Submerged epithelial cultures will be established at each visit to the clinic and assays described above carried out within 2 weeks to determine effects of triheptanoin treatment on cell death, mitochondrial function and signalling. The primary outcome variable will be percent cell death induced by glucose deprivation in cell culture.

SECONDARY OUTCOMES:
Scales for assessment and rating of ataxia | Day 1, Day 120, Day 240, Day 360
  Scales for assessment and rating of ataxia is a validated cerebellar ataxia tool, measuring gait (scale 0-8), stance (scale 0-6), sitting (scale 0-4), speech (scale 0-6), finger-chase test scale 0-4), finger nose-test (scale 0-4), fast alternating movements (scale 0-4) and heel-shin test (scale 0-4). 0 indicates normal function, escalating numbers in the scale domains indicate increased difficultly with the measured tasks.
International Cooperative Ataxia Rating Scale | Day 1, Day 120, Day 240, Day 360
  International Cooperative Ataxia Rating Scale is a scale recorded out of 100 with 19 items and 4 sub-scales and has been used in A-T. 0 indicates normal function, escalating numbers in the scale domains indicate increased difficulty with the measured tasks.
Speech Pathology Assessments | Day 1, Day 120, Day 240, Day 360
  Speech perception and intelligibility will be defined using a standardised instrument.
Ophthalmology assessments | Day 1, Day 120, Day 240, Day 360
  The EyeSeeCam system will acquire calibrated recordings and quantified analysis of eye movements for assessment of saccadic latency, fixation stability, optokinetic nystagmus and vestibulo-ocular reflex response, and ocular coherence tomography scans provide detailed images of retinal nerve fibre layer.
MRI lung imaging | Performed at Day 1 and Day 360 in suitable participants
  MRI with ultra-short echo time sequences including Pointwise Encoding Time Reduction with Radial Acquisition and Volumetric Interpolated Breath-hold Examination will define lung structure, and diffusion weighted imaging to estimate inflammatory lung changes.
Spirometry Vital capacity (litres) | Day 1, Day 120, Day 240, Day 360
  Lung function will be measured using conventional spirometry in those able to perform the test.
Spirometry Forced vital capacity (litres) | Day 1, Day 120, Day 240, Day 360
  Lung function will be measured using conventional spirometry in those able to perform the test.
Spirometry Forced expiratory volume in one second (litres) | Day 1, Day 120, Day 240, Day 360
  Lung function will be measured using conventional spirometry in those able to perform the test.
Spirometry Peak expiratory flow (L.min-1) | Day 1, Day 120, Day 240, Day 360
  Lung function will be measured using conventional spirometry in those able to perform the test.
Upper respiratory microbiome | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  DNA extraction and sequencing via Qiagen DNA isolation kit then 16S rRNA sequencing16S rRNA sequencing
Faecal microbiome | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  DNA extraction and sequencing via Qiagen DNA isolation kit then 16S rRNA sequencing16S rRNA sequencing to identify faecal microbial composition. 1D 1H NMR spectroscopy and gas chromatography for short chain fatty acids and other metabolites.
Intestinal permeability | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  Lipopolysaccharide, Lipopolysaccharide binding protein and Zonulin analys by standard ELISA assays.

OTHER OUTCOMES:
Survival and inflammatory phenotype of airway epithelial cells, macrophages and in serum | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  Pro-inflammatory cytokines IL-8 (g/ml) and TNF-α (g/ml) and a decreased level of the inflammasome dependent cytokine IL-β (g/ml) will be assayed in the supernatants of epithelial cell cultures and macrophages and in serum. All will be quantitated via AlphaLISA according to the manufacturers' protocol (Perkin Elmer, MA, USA).
Serum metabolomic biomarker | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  SWATH-MS based methods to identify candidate small molecule biomarkers in participants validated against an independent study cohort. Small molecules will be enriched from serum by organic solvent precipitation of proteins followed by solid phase extraction and/or filtration.
Air Displacement Plethysmography | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  The BOD POD is the device used to measure body volume giving reliable and reproducible results to determine fat mass and lean body mass. The BOD POD is quick, safe, non-invasive and able to be used in both the adult and paediatric population
Quality of Life Measures | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  Paediatric Side Effect Questionnaire is a 19-item measure consisting of five sub-scales: cognitive (six items), motor (four items), behavioural (three items), general neurological (four items), and weight (two items) side effects. The investigators will add five items for gastrointestinal side effects to the questionnaire, including gastrointestinal pain, acid reflux, vomiting, diarrhoea, and constipation. The scale will be recorded from 0 to 96. 0 indicates normal function, escalating numbers in the scale domains indicate increased difficultly with the measured task.
Neurofilament light chain | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  Neurofilament light chain will be quantified using the single-molecule (Simoa) array method and the Simoa NF-light assay (Quanterix, MA, US) on an HD-1platform (GBIO).
Nutritional assessments | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  Standardised tool used include, validated diet history tools such as simplified nutritional appetite questionnaire, and weight and height.
body mass index in kg/m^2 | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  weight (kg) / [height (m)]2
Resting energy expenditure | Day 1, Day 60, Day 120, Day 180, Day 240, Day 300, Day 360
  Resting energy expenditure will be calculated using the Harris-Benedict Equations (calories/day):
  Male: (66.5 + 13.8 X weight) + (5.0 X height) - (6.8 X age) Female: (665.1 + 9.6 X weight) + (1.8 X height) - (4.7 X age) weight in kilograms, height in centimeters, age in years
Seamless Phase II to Phase III go/no-go criteria | Interim independent data safety management committee analysis Day 180 and Day 240
  The A-T2020/01 standing platform trial provides a resource to enable a promising therapy for AT to be rapidly evaluated and to facilitate seamless transition from a Phase II to a Phase III study. Initially the platform will support a phase IIA/IIB study, but if the new intervention being evaluated is considered effective then we plan to move seamlessly from this Phase IIA/IIB study to a Phase III. The move to a Phase III trial will be guided by a pre-defined threshold for the probability of a successful intervention during phase III, which will be established in planning the Phase IIA/IIB trial and agreed by regulatory authorities for pivotal studies. If a seamless transition to Phase III is considered feasible, the trial investigators and the trial statistics team will provide the iDSMB and TSC with a Phase III proposal, and if this was approved by the iDSMB and TSC then further recruitment to the target number determined would be undertaken.

CONTACTS AND LOCATIONS:
Overall Officials: David Coman, MBBS FRACP, Principal Investigator — Queensland Children's Hospital
Locations (1):
- Queensland Children's Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Z, Kozlov S, Lavin MF, Person MD, Paull TT. ATM activation by oxidative stress. Science. 2010 Oct 22;330(6003):517-21. doi: 10.1126/science.1192912. PMID 20966255
- [Result] Zannolli R, Buoni S, Betti G, Salvucci S, Plebani A, Soresina A, Pietrogrande MC, Martino S, Leuzzi V, Finocchi A, Micheli R, Rossi LN, Brusco A, Misiani F, Fois A, Hayek J, Kelly C, Chessa L. A randomized trial of oral betamethasone to reduce ataxia symptoms in ataxia telangiectasia. Mov Disord. 2012 Sep 1;27(10):1312-6. doi: 10.1002/mds.25126. Epub 2012 Aug 23. PMID 22927201
- [Result] Gueven N, Luff J, Peng C, Hosokawa K, Bottle SE, Lavin MF. Dramatic extension of tumor latency and correction of neurobehavioral phenotype in Atm-mutant mice with a nitroxide antioxidant. Free Radic Biol Med. 2006 Sep 15;41(6):992-1000. doi: 10.1016/j.freeradbiomed.2006.06.018. Epub 2006 Jul 4. PMID 16934683
- [Result] Valentin-Vega YA, Maclean KH, Tait-Mulder J, Milasta S, Steeves M, Dorsey FC, Cleveland JL, Green DR, Kastan MB. Mitochondrial dysfunction in ataxia-telangiectasia. Blood. 2012 Feb 9;119(6):1490-500. doi: 10.1182/blood-2011-08-373639. Epub 2011 Dec 5. PMID 22144182
- [Result] Gillingham MB, Heitner SB, Martin J, Rose S, Goldstein A, El-Gharbawy AH, Deward S, Lasarev MR, Pollaro J, DeLany JP, Burchill LJ, Goodpaster B, Shoemaker J, Matern D, Harding CO, Vockley J. Triheptanoin versus trioctanoin for long-chain fatty acid oxidation disorders: a double blinded, randomized controlled trial. J Inherit Metab Dis. 2017 Nov;40(6):831-843. doi: 10.1007/s10545-017-0085-8. Epub 2017 Sep 4. PMID 28871440
- [Result] Roe CR, Brunengraber H. Anaplerotic treatment of long-chain fat oxidation disorders with triheptanoin: Review of 15 years Experience. Mol Genet Metab. 2015 Dec;116(4):260-8. doi: 10.1016/j.ymgme.2015.10.005. Epub 2015 Oct 24. PMID 26547562
- [Result] Roe CR, Mochel F. Anaplerotic diet therapy in inherited metabolic disease: therapeutic potential. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):332-40. doi: 10.1007/s10545-006-0290-3. PMID 16763896
- [Result] Schiffmann R, Wallace ME, Rinaldi D, Ledoux I, Luton MP, Coleman S, Akman HO, Martin K, Hogrel JY, Blankenship D, Turner J, Mochel F. A double-blind, placebo-controlled trial of triheptanoin in adult polyglucosan body disease and open-label, long-term outcome. J Inherit Metab Dis. 2018 Sep;41(5):877-883. doi: 10.1007/s10545-017-0103-x. Epub 2017 Nov 6. PMID 29110179
- [Result] Hainque E, Caillet S, Leroy S, Flamand-Roze C, Adanyeguh I, Charbonnier-Beaupel F, Retail M, Le Toullec B, Atencio M, Rivaud-Pechoux S, Brochard V, Habarou F, Ottolenghi C, Cormier F, Meneret A, Ruiz M, Doulazmi M, Roubergue A, Corvol JC, Vidailhet M, Mochel F, Roze E. A randomized, controlled, double-blind, crossover trial of triheptanoin in alternating hemiplegia of childhood. Orphanet J Rare Dis. 2017 Oct 2;12(1):160. doi: 10.1186/s13023-017-0713-2. PMID 28969699
- [Result] Hainque E, Gras D, Meneret A, Atencio M, Luton MP, Barbier M, Doulazmi M, Habarou F, Ottolenghi C, Roze E, Mochel F. Long-term follow-up in an open-label trial of triheptanoin in GLUT1 deficiency syndrome: a sustained dramatic effect. J Neurol Neurosurg Psychiatry. 2019 Nov;90(11):1291-1293. doi: 10.1136/jnnp-2018-320283. Epub 2019 Apr 4. No abstract available. PMID 30948626
- [Result] Hadera MG, Smeland OB, McDonald TS, Tan KN, Sonnewald U, Borges K. Triheptanoin partially restores levels of tricarboxylic acid cycle intermediates in the mouse pilocarpine model of epilepsy. J Neurochem. 2014 Apr;129(1):107-19. doi: 10.1111/jnc.12610. Epub 2013 Dec 2. PMID 24236946
- [Result] Hadera MG, McDonald T, Smeland OB, Meisingset TW, Eloqayli H, Jaradat S, Borges K, Sonnewald U. Modification of Astrocyte Metabolism as an Approach to the Treatment of Epilepsy: Triheptanoin and Acetyl-L-Carnitine. Neurochem Res. 2016 Feb;41(1-2):86-95. doi: 10.1007/s11064-015-1728-5. Epub 2015 Oct 3. PMID 26433381
- [Result] Yeo AJ, Henningham A, Fantino E, Galbraith S, Krause L, Wainwright CE, Sly PD, Lavin MF. Increased susceptibility of airway epithelial cells from ataxia-telangiectasia to S. pneumoniae infection due to oxidative damage and impaired innate immunity. Sci Rep. 2019 Feb 22;9(1):2627. doi: 10.1038/s41598-019-38901-3. PMID 30796268
- [Result] McGrath-Morrow SA, Collaco JM, Detrick B, Lederman HM. Serum Interleukin-6 Levels and Pulmonary Function in Ataxia-Telangiectasia. J Pediatr. 2016 Apr;171:256-61.e1. doi: 10.1016/j.jpeds.2016.01.002. Epub 2016 Feb 2. PMID 26851119
- [Result] McGrath-Morrow SA, Ndeh R, Collaco JM, Rothblum-Oviatt C, Wright J, O'Reilly MA, Singer BD, Lederman HM. Inflammation and transcriptional responses of peripheral blood mononuclear cells in classic ataxia telangiectasia. PLoS One. 2018 Dec 26;13(12):e0209496. doi: 10.1371/journal.pone.0209496. eCollection 2018. PMID 30586396
- [Result] Ross LJ, Capra S, Baguley B, Sinclair K, Munro K, Lewindon P, Lavin M. Nutritional status of patients with ataxia-telangiectasia: A case for early and ongoing nutrition support and intervention. J Paediatr Child Health. 2015 Aug;51(8):802-7. doi: 10.1111/jpc.12828. Epub 2015 Feb 6. PMID 25656498
- [Result] Morita DA, Glauser TA, Modi AC. Development and validation of the Pediatric Epilepsy Side Effects Questionnaire. Neurology. 2012 Sep 18;79(12):1252-8. doi: 10.1212/WNL.0b013e3182635b87. Epub 2012 Aug 8. PMID 22875082
- [Result] Yeo AJ, Chong KL, Gatei M, Zou D, Stewart R, Withey S, Wolvetang E, Parton RG, Brown AD, Kastan MB, Coman D, Lavin MF. Impaired endoplasmic reticulum-mitochondrial signaling in ataxia-telangiectasia. iScience. 2020 Dec 23;24(1):101972. doi: 10.1016/j.isci.2020.101972. eCollection 2021 Jan 22. PMID 33437944